CLINICAL TRIAL: NCT06471699
Title: A Randomized Trial of the Effect of Continuous Glucose Monitoring (CGM) in Individuals With Newly Diagnosed Type 2 Diabetes
Brief Title: The Effect of Continuous Glucose Monitoring in Individuals With Newly Diagnosed Type 2 Diabetes
Acronym: CHANGE-diab
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: The Swedish Research Council (Other Government); Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 282418
Record Dates: First submitted 2024-06-11; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continous Glucose Monitoring (Experimental): Participants will be randomized to intervention Continous Glucose Monitoring (CGM)
  Interventions: Device: Continous Glucose Monitoring
- Self Monitoring Blood Glucose (Active Comparator): Participants will be randomized to control Self Monitoring Blood Glucose (SMBG)
  Interventions: Other: Self monitoring blood glucose

INTERVENTIONS:
Device: Continous Glucose Monitoring — The aim is to examine if the use of CGM will give the participants a significant support to implement lifestyle improvements in individuals with new on-set type 2 diabetes
  Arms: Continous Glucose Monitoring
Other: Self monitoring blood glucose — Capillary testing as in standard procedure
  Arms: Self Monitoring Blood Glucose

SUMMARY:
The aim of the current study is to evaluate effectiveness, sustainability and satisfaction of CGM in adult persons with newly diagnosed type 2 diabetes. The study is a randomized clinical trial randomizing patients to CGM or SMBG over 26 weeks with a follow-up period up to 70 weeks. An extension period will exist between 26 and 70 weeks. Between 26-52 weeks both groups will use only capillary testing for glucose monitoring and during 53-70 weeks the group initially randomized to capillary testing will use CGM. During the extension period similar variables will be evaluated as during the main phase of the trial including HbA1c, CGM-metrics, glucose-lowering medications, physical activity, treatment satisfaction and well-being.

DETAILED DESCRIPTION:
A keystone in preventing complications in persons with type 2 diabetes is good glycaemic control as soon as possible after onset of diabetes. The basic treatment is optimizing lifestyle factors with increased physical activity, weight control and a healthy diet. In addition to glucose control, it is important that blood pressure and blood lipids are well regulated. Self-monitoring of blood glucose (SMBG) by repeated capillary glucose measurements has been a standard for regulating plasma glucose levels and to give information about the influence of lifestyle. In recent years continuous glucose monitoring (CGM) has become an option for guiding the patient by immediate feedback on the influence of lifestyle, such as physical activity and diet.

Previous studies indicate that CGM helps and encourages people with type 2 diabetes to improve their lifestyle and that it is highly appreciated.. However, it is relatively expensive and the effect of CGM on glycaemic control may fade over time.

No previous study has examined the effect of CGM on lifestyle in individuals with newly diagnosed type 2 diabetes. Individuals with newly diagnosed diabetes are more prone to change their lifestyle while quick improvement of glucose measurements also is of uttermost importance.

The aim of the current study is to evaluate effectiveness, sustainability and satisfaction of CGM in adult persons with newly diagnosed type 2 diabetes. The study is a randomized clinical trial randomizing patients to CGM or SMBG over 26 weeks with a follow-up period up to 70 weeks. The primary endpoint is effect on HbA1c over 26 weeks. Other essential endpoints over 26 weeks of treatment include effects on time in range, glucose variability, treatment satisfaction, well-being and weight over 26 weeks of treatment. Need of adding glucose lowering medications will also be compared between the treatment groups. An extension period will exist between 26 and 70 weeks. Between 26-52 weeks both groups will use only capillary testing for glucose monitoring and during 53-70 weeks the group initially randomized to capillary testing will use CGM. During the extension period similar variables will be evaluated as during the main phase of the trial including HbA1c, CGM-metrics, glucose-lowering medications, physical activity, treatment satisfaction and well-being.

In total 238 patients will be included in this study, carried out at 30 health care centres in Sweden

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. Adults 18 years or older
3. Written Informed Consent
4. HbA1c greater than or equal to 58 mmol/mol (7.5% DCCT standard) and less than 100 mmol/mol
5. Type 2 diabetes diagnosis <4 weeks
6. Body mass index > 25 kg/m2

Exclusion Criteria:

1. Pregnancy or planned pregnancy for the study duration
2. Type 1 diabetes
3. Judged to be in need of insulin
4. Severe cognitive dysfunction or other disease, which is judged by the physician to be not suitable for inclusion.
5. History of allergic reaction to chlorhexidine or alcohol anti-septic solution.
6. Abnormal skin at the anticipated glucose sensor attachment sites (excessive hair, burn, inflammation, infection, rash, and/or tattoo).
7. Participation in another study.
8. Other investigator-determined criteria unsuitable for patient participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 6 months
  Differences in changes in HbA1c between the CGM and SMBG group.

SECONDARY OUTCOMES:
Time in range (TIR) | 6 months, 52 and 70 weeks
  Differences in changes Time in range (TIR) over 26 weeks of treatment measured by CGM between the CGM and SMBG group.
Glucose variability | 6 months, 52 and 70 weeks
  Differences in changes in Glucose variability over 26 weeks of treatment measured by CGM between the CGM and SMBG group.
Treatment satisfaction | 6 months, 52 and 70 weeks
  Differences in changes in treatment satisfaction over 26 weeks of treatment measured by validated questionnaires between the CGM and SMBG group. Treatment satisfaction measured with the questionnaires DTSQs (Diabetes Treatment Satisfaction Questionnaire, 0-48 points with best treatment 48p) and DTSQc follow-up (-24 to 24 points with best treatment 24P)
Well-being | 6 months, 52 and 70 weeks
  Differences in changes in well-being over 26 weeks of treatment measured by validated questionnaires between the CGM and SMBG group. Wellbeing will be measured with the questionnaires WHO5 (World Health Organisation, 0-25points with the best wellbeing 25P).
Weight | 6 months, 52 and 70 weeks
  Differences in changes in weight over 26 weeks of treatment between the CGM and SMBG group.

OTHER OUTCOMES:
Physical activity | 26,52 och 70 weeks
  Exploratory objectives - differences in changes in physical activity measured with a questionnaire with self-reported data, IPAC (International Physical Activity Questionnaire, Physical activity estimated through transforming the answers about physical activity into METs with the highest METs as the most physicallay active) between the CGM and SMBG group.
Waist circumference | 26,52 och 70 weeks
  Exploratory objectives - differences in changes in waist circumference between the CGM and SMBG group.
Fasting glucose | 26,52 och 70 weeks
  Exploratory objectives - differences in changes in fasting glucose between the CGM and SMBG group.
Blood pressure | 26,52 och 70 weeks
  Exploratory objectives - differences in changes in blood pressure, both systolic and diastolic, between the CGM and SMBG group.
Triglycerides | 26,52 och 70 weeks
  Exploratory objectives - differences in changes in triglycerides between the CGM and SMBG group.
Reduction of HbA1c | 26,52 och 70 weeks
  Differences in changes of HbA1c by 5 mmol/mol (0.5% in DCCT) or more between the CGM and the SMBG group.
Reduction of HbA1c | 26,52 och 70 weeks
  Differences in changes of HbA1c by 10 mmol/mol (0.5% in DCCT) or more between the CGM and the SMBG group.
Time in high glucose levels | 26,52 och 70 weeks
  Differences in time of high glucose levels as measured by CGM (above 10.0 mmol/l and above 13.9 mmol/l) between the CGM and the SMBG group